CLINICAL TRIAL: NCT00574444
Title: Laparoscopic Assisted Transvaginal Endoscopic Diagnostic Peritoneoscopy in Women With Pelvic Pain
Brief Title: Transvaginal Diagnostic Study in Women With Pelvic Pain
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator moved to another institution.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1096837
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Pelvic Pain
Keywords: transvaginal peritoneoscopy
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Procedure (Experimental): Procedure/Surgery: transvaginal diagnostic peritoneoscopy For patients with pelvic pain, a transvaginal procedure can be done to explore the abdomen. Entering through the vagina, will hopefully decrease the number of ports in the abdomen and decrease pain and healing time.
  Interventions: Procedure: transvaginal diagnostic peritoneoscopy

INTERVENTIONS:
Procedure: transvaginal diagnostic peritoneoscopy — For patients with pelvic pain, a transvaginal procedure can be done to explore the abdomen. Entering through the vagina, will hopefully decrease the number of ports in the abdomen and decrease pain and healing time.

SUMMARY:
We propose a phase I study of laparoscopic assisted, transvaginal peritoneoscopy by using flexible endoscopy in female patients with pelvic pain. It is designed as a hybrid procedure with laparoscopy using one port for adequate safety with the ultimate goal in the future that transvaginal NOTES can replace therapeutic pelviscopy for this indication. The standard number of port sites for diagnostic laparoscopy is 2-3. By reducing the number and size of laparoscopic port, patients should already experience benefits from this hybrid procedure.

DETAILED DESCRIPTION:
Approximately 50% of patients with chronic pelvic pain will have a normal laparoscopy. The vast majority of women with endometriosis, chronic pelvic pain and absence of ovarian endometriomata determined by ultrasound will have revised ASRM Stage I or II (peritoneal) disease with preservation of the posterior cul-de-sac. This sparing of the posterior cul-de-sac may offer a preferable route of entry for endoscopic surgery compared to the current standard of care.

Despite all the advantages of laparoscopic surgery, it is not free of risks and pain, and creates scars, which themselves are associated with complications such as abdominal wall hernias and adhesions.

Within this scenario, a new surgical procedure has emerged, called natural orifice transluminal endoscopic surgery (NOTES). This technique uses existing orifices of the body for introducing optical systems and surgical instruments into the peritoneal cavity by avoiding penetration of the abdominal wall. The expectations are no postoperative pain, optimal cosmesis without any visable scars and shorter recovery similar to therapeutic endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 and older who have an indication and scheduled for laparoscopic peritoneoscopy.

Exclusion Criteria:

* Known pelvic adhesive disease or greater than stage II endometriosis or sonographic evidence of endometrioma.
* BMI over 30.
* Major comorbidities - including diabetes, myocardial infarction, congestive heart failure, stroke, history of cancer or currently undergoing chemotherapy, autoimmune disease requiring immunosuppressive or steroid therapy .
* Any primary bowel disease (IBD, sprue, obstruction, acute appendicitis, gastric bypass, etc.).
* Pregnancy.
* Any known PID, tuboovarian mass or abscess, or active sexually transmitted infection.
* Retroflexed uterus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety and feasibility of the procedure. | by January 2010

SECONDARY OUTCOMES:
Measurement of patient's post operative pain | post-operative day 1 and post-operative day 7

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Thaler, MD, Principal Investigator — Dept. of General Surgery at UMHC
Locations (1):
- University of Missouri Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No